CLINICAL TRIAL: NCT04044664
Title: A Study to Evaluate the Safety and Efficacy of NYX-783 in Subjects With Post-Traumatic Stress Disorder
Brief Title: Safety and Efficacy of NYX-783 in Subjects With Post-Traumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aptinyx (Industry)
Collaborators: Premier Research (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NYX-783-2004
Record Dates: First submitted 2019-07-09; First posted 2019-08-05 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive placebo or NYX-783.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule
- NYX-783 Low Dose (10 mg QD) (Experimental)
  Interventions: Drug: NYX-783
- NYX-783 High Dose (50 mg QD) (Experimental)
  Interventions: Drug: NYX-783

INTERVENTIONS:
Drug: Placebo oral capsule — Matching placebo capsules.
  Arms: Placebo
Drug: NYX-783 — NYX-783 is a small molecule that modulates the N-methyl-D-aspartate receptor (NMDAR).
  Arms: NYX-783 High Dose (50 mg QD); NYX-783 Low Dose (10 mg QD)

SUMMARY:
To evaluate the safety, tolerability, and response profile of NYX-783 in a Post-Traumatic Stress Disorder population.

DETAILED DESCRIPTION:
The study will be a 10 to 12-week study, including a 1 to 3-week screening Period, followed by a double-blind, randomized, placebo-controlled, parallel-group Treatment Period, and a 1-week follow-up Period. Subjects eligible for the study will be randomized to receive either NYX-783 (4-weeks) or placebo (4 or 8-weeks).

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of PTSD [Post Traumatic Stress Disorder, according to DSM-5 (Diagnostic and Statistical Manual of Mental Disorders)] with the primary traumatic event occurring ≥12 months prior to screening.
* PCL-5 (PTSD Checklist for DSM-5) ≥38 at screening.
* CAPS-5 (Clinician-Administered PTSD Scale for DSM-5) total score ≥30 at screening.

Exclusion Criteria:

* Complex PTSD.
* Trauma focused psychotherapies.
* Primary traumatic event occurred prior to 2001.
* Primary traumatic event was followed by further major traumatic life episodes.
* Other psychiatric disorders that is the primary focus of treatment or followed/worsened since exposure to the trauma (except for major depressive disorder or anxiety disorders that followed exposure to the trauma or an anxiety disorder that showed a worsening after trauma)
* Current use of medications with primarily central nervous system activities
* Other clinically significant medical histories that may interfere with completing the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (37):
  - Aptinyx Clinical Site, Tuscaloosa, Alabama
  - Aptinyx Clinical Site, Phoenix, Arizona
  - Aptinyx Clinical Site, Little Rock, Arkansas
  - Aptinyx Clinical Site, Bellflower, California
  - Aptinyx Clinical Site, Glendale, California
  - Aptinyx Clinical Site, Imperial, California
  - Aptinyx Clinical Site, Oakland, California
  - Aptinyx Clinical Site, Oceanside, California
  - Aptinyx Clinical Site, Orange, California
  - Aptinyx Clinical Site, Riverside, California
  - Aptinyx Clinical Site, San Diego, California
  - Aptinyx Clinical Site, San Marcos, California
  - Aptinyx Clinical Site, Santa Ana, California
  - Aptinyx Clinical Site, Temecula, California
  - Aptinyx Clinical Site, Torrance, California
  - Aptinyx Clinical Site, Colorado Springs, Colorado
  - Aptinyx Clinical Site, Norwich, Connecticut
  - Aptinyx Clinical Site, Jacksonville, Florida
  - Aptinyx Clinical Site, Lauderhill, Florida
  - Aptinyx Clinical Site, Orlando, Florida
  - Aptinyx, Atlanta, Georgia
  - Aptinyx Clinical Site, Atlanta, Georgia
  - Aptinyx Clinical Site, Hoffman Estates, Illinois
  - Aptinyx Clinical Site, Boston, Massachusetts
  - Aptinyx Clinical Site, Las Vegas, Nevada
  - Aptinyx Clinical Site, Berlin, New Jersey
  - Aptinyx Clinical Site, Cedarhurst, New York
  - Aptinyx Clinical Site, New York, New York
  - Aptinyx Clinical Site, Staten Island, New York
  - Aptinyx Clinical Site, Salisbury, North Carolina
  - Aptinyx Clinical Site, Canton, Ohio
  - Aptinyx Clinical Site, Cincinnati, Ohio
  - Aptinyx Clinical Site, Oklahoma City, Oklahoma
  - Aptinyx Clinical Site, Memphis, Tennessee
  - Aptinyx Clinical Site, Austin, Texas
  - Aptinyx Clinical Site, San Antonio, Texas
  - Aptinyx Clinical Site, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to Placebo, NYX-783 50mg QD, or NYX-783 10mg QD during Stage 1. Participants were re-randomized to Placebo, NYX-783 50mg QD, or NYX-783 10mg QD in Stage 2. Participants who received Placebo in Stage 1 were classified as Responders or Non-responders in Stage 2.
  160 subjects were randomized. 7 subjects received 50mg QW in a prior protocol version; they were not assigned to the Arms/Groups above. 1 subject was randomized in Stage 1 but did not receive study drug.
Period: Stage 1
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD)
Started | 103 | 26 | 23
Completed | 86 | 19 | 20
Not Completed | 17 | 7 | 3
Not completed — Adverse Event | 3 | 3 | 1
Not completed — Lost to Follow-up | 3 | 2 | 2
Not completed — Withdrawal by Subject | 9 | 1 | 0
Not completed — noncompliance, personal reason | 2 | 0 | 0
Not completed — randomization error | 0 | 1 | 0
Period: Stage 2
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD)
Started | 76 | 26 | 22
From Placebo, Responder | 20 | 13 | 11
From Placebo, Non-Responder | 18 | 13 | 11
From NYX-783 (10 mg or 50 mg) | 38 | 0 | 0
Completed | 67 | 24 | 21
Not Completed | 9 | 2 | 1
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — protocol deviation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD) | Total
Number analyzed (Participants) | 103 | 26 | 23 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (11.42) | 43.8 (12.54) | 43.7 (11.96) | 41.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 15 | 16 | 92
  Male | 42 | 11 | 7 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 4 | 0 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 23 | 6 | 6 | 35
  White | 75 | 17 | 15 | 107
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 103 | 26 | 23 | 152
Baseline CAPS-5 Total Score [Mean (Standard Deviation); unit: units on a scale] — CAPS-5 [Clinician Administered PTSD Scale for DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition)] is a structured interview for diagnosis and assessment of PTSD. The assessor combines information about frequency and intensity of an item into a severity rating (0-4). CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms (minimum score 0, maximum score 80). A higher score corresponds to more severe PTSD.
  units on a scale | 40.6 (7.58) | 36.5 (7.37) | 38.3 (8.26) | 39.6 (7.76)

OUTCOME MEASURES:

1. Primary Outcome: CAPS-5 [Clinician-Administered PTSD Scale for DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition)] Total Score and Subscores
Description: CAPS-5 [Clinician Administered PTSD Scale for DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition)] is a structured interview for diagnosis and assessment of PTSD. The assessor combines information about frequency and intensity of an item into a severity rating (0-4). CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: intrusions (items 1-5, minimum score 0, maximum score 20), avoidance (items 6-7, minimum score 0, maximum score 8), negative alterations in cognitions and mood (items 8-14, minimum score 0, maximum score 28), and alterations in arousal and reactivity (items 15-20, minimum score 0, maximum score 24). CAPS-5 Total Scores range from 0 to 80. A higher score corresponds to more severe PTSD.
Time Frame: Change from baseline to week 4 (Stage 1)
Population: Intent to Treat, all randomized subjects
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD)
Number analyzed (Participants) | 103 | 26 | 23
units on a scale
  CAPS-5 Total Score | -13.4 (1.06) | -15.7 (2.24) | -11.6 (2.19)
  Intrusion sub-score | -4.4 (0.35) | -4.3 (0.75) | -3.7 (0.72)
  Avoidance sub-score | -1.8 (0.21) | -2.2 (0.44) | -1.4 (0.44)
  Cognition and Mood sub-score | -4.2 (0.5) | -5.7 (1.05) | -3.4 (1.04)
  Arousal and Reactivity sub-score | -2.7 (.28) | -4.1 (0.61) | -3.5 (0.59)
Statistical Analysis 1: Comparison: Placebo vs NYX-783 High Dose (50 mg QD); CAPS-5 Total Score; Test type: Other; p = 0.1728, t-test, 1 sided
Statistical Analysis 2: Comparison: Placebo vs NYX-783 High Dose (50 mg QD); Cognition and Mood sub-score; Test type: Other; p = 0.0962, t-test, 1 sided
Statistical Analysis 3: Comparison: Placebo vs NYX-783 High Dose (50 mg QD); Arousal and Reactivity sub-score; Test type: Other; p = 0.0191, t-test, 1 sided

2. Secondary Outcome: PCL-5 (PTSD-Checklist for DSM-5)
Description: Assess the effect of NYX-783 compared to placebo in changes of symptoms as measured by PCL-5. The PCL-5 ranges from 0 to 80; a higher score corresponds to more severe PTSD.
Time Frame: Change from baseline to week 4 (Stage 1)
Population: Intent to Treat, all randomized subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD)
Number analyzed (Participants) | 103 | 26 | 23
units on a scale | -16.6 (14.75) | -19.9 (13.58) | -17.0 (16.45)

3. Secondary Outcome: PSQI (Pittsburgh Sleep Quality Index) Global Score
Description: Assess the effects of NYX-783 compared to placebo in changes in sleep quality as measure by the PSQI Global Score. The PSQI is a questionnaire to assess sleep quality and disturbances. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. A score >5 indicates significant sleep disturbance.
Time Frame: Change from baseline to week 4 (Stage 1)
Population: Intent to Treat, all randomized subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD)
Number analyzed (Participants) | 103 | 26 | 23
units on a scale | -1.5 (3.37) | -1.2 (2.89) | -1.8 (4.04)

4. Secondary Outcome: PSQI-A (Pittsburgh Sleep Quality Index-Addendum) Global Score
Description: Assess the effects of NYX-783 compared to placebo in changes in sleep quality as measure by the PSQI-A Global Score. The PSQI-A score ranges from 0-21; lower scores represent less disruptive behavior.
Time Frame: Change from baseline to week 4 (Stage 1)
Population: Intent to Treat, all randomized subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD)
Number analyzed (Participants) | 86 | 19 | 20
units on a scale | -2.9 (3.76) | -1.9 (2.66) | -3.1 (4.84)

5. Secondary Outcome: BAC (Brief Assessment of Cognition) Symbol Coding
Description: Assess the effect of NYX-783 compared to placebo in changes in cognitive function as measured by the BAC Symbol Coding. BAC symbol coding score is a count which ranges from 0 to 110; higher scores represent higher function.
Time Frame: Change from baseline to week 4 (Stage 1)
Population: Intent to Treat, all randomized subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD)
Number analyzed (Participants) | 103 | 26 | 23
units on a scale | 3.8 (8.07) | 2.9 (9.00) | 1.3 (5.37)

6. Secondary Outcome: CGI-S (Clinical Global Impression - Severity)
Description: Assess the effect of NYX-783 compared to placebo in the change in global clinical severity of PTSD symptoms as measured by the CGI-S. The Clinical Global Impressions-Severity (CGI-S) score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill subjects).
Time Frame: Change from baseline to week 4 (Stage 1)
Population: Intent to Treat, all randomized subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD)
Number analyzed (Participants) | 103 | 26 | 23
units on a scale | -1.1 (1.09) | -1.2 (1.03) | -1.3 (0.99)

7. Secondary Outcome: HADS-A (Hospital Anxiety and Depression Scale)
Description: The HADS is a self-assessment tool consisting of two subscales, one for anxiety (HADS-A) and one for depression (HADS-D). Scores for items in each subscale of the HADS are summed to produce an anxiety score (HADS-A) or a Depression score (HADS-D), or can be added to produce a total score (HADS-T). Each item is rated on a 4-point scale (ranging from 0 = no not at all, to 3 = yes definitely), for a total score ranging from 0-42 and sub scores for anxiety or depression ranging from 0-21 for each subscale. Higher scores represent more severe anxiety or depression. HADS-A is presented here.
Time Frame: From baseline to week 4 (Stage 1)
Population: Intent to Treat, all randomized subjects
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD)
Number analyzed (Participants) | 103 | 26 | 23
units on a scale | -3.0 (.34) | -4.4 (0.72) | -4.2 (0.7)
Statistical Analysis 1: Comparison: Placebo vs NYX-783 High Dose (50 mg QD); Test type: Other; p = 0.0452, t-test, 1 sided
Statistical Analysis 2: Comparison: Placebo vs NYX-783 Low Dose (10 mg QD); Test type: Other; p = 0.0614, t-test, 1 sided

8. Post Hoc Outcome: Responders (30% and 50% Improvement From Baseline) in CAPS-5 Total Score
Description: Clinician Administered PTSD Scale for DSM-5 (CAPS-5) is a 30-item structured interview for diagnosis and assessment of PTSD. A higher score corresponds to more severe PTSD.
Time Frame: Baseline to Week 4 (Stage 1)
Population: Intent to Treat, subjects who completed Week 4
Measure: Number; unit: participants
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD)
Number analyzed (Participants) | 103 | 26 | 23
participants
  30% decrease from baseline | 38 | 14 | 9
  50% decrease from baseline | 23 | 9 | 6
Statistical Analysis 1: Comparison: Placebo vs NYX-783 High Dose (50 mg QD); greater than or equal to 30% decrease from baseline; Test type: Other; p = 0.0182, t-test, 1 sided
Statistical Analysis 2: Comparison: Placebo vs NYX-783 High Dose (50 mg QD); greater than or equal to 50% decrease from baseline; Test type: Other; p = 0.0705, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Stage 1: 4 weeks, Stage 2: 4 weeks
Description: Adverse Events were assessed at protocol specified study visits.
Arm/Group | Placebo | NYX-783 High Dose (50 mg QD) | NYX-783 Low Dose (10 mg QD)
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/52 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/52 | 0/46
Other Adverse Events (participants affected / at risk) | 9/141 | 4/52 | 3/46
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=141) | NYX-783 High Dose (50 mg QD) (N=52) | NYX-783 Low Dose (10 mg QD) (N=46)
Headache (Nervous system disorders) | 8 (8) | 2 (2) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT04044664/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT04044664/SAP_001.pdf